CLINICAL TRIAL: NCT00126217
Title: BCG Vaccination and Childhood Morbidity and Mortality: Interventions With Possible Implications for the Immunisation Policy in Developing Countries. Revaccination of Young Children With BCG Vaccine.
Brief Title: Revaccination of Young Children With Bacille Calmette Guerin (BCG) Vaccine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: A cluster of deaths in the BCG-arm compared with controls
Sponsor: Bandim Health Project (Other)
Collaborators: International Cooperation with Developing Countries (Other); Leiden University Medical Centre, DEPT of Parasitology, Leiden Holland (Other); Medical Research Council Unit, The Gambia (Other)
Responsible Party: Peter Aaby, Professor, Apartado 861, Bissau,Guinea-Bissau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICA4-CT-2002-10053-REVAC; EU contract ICA4-CT-2002-10053
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Malaria
Keywords: Non-specific effects of vaccines; Infant mortality; Morbidity; Low income country; Malaria; BCG; immunisation; BCG revaccination; Tuberculin; Mortality
MeSH Terms: conditions — Malaria; Infant Death

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Bacille Calmette Guerin (BCG)
- 2 (No Intervention)

INTERVENTIONS:
Biological: Bacille Calmette Guerin (BCG) — 0,1 ml, revaccination at 19 months of age
  Arms: 1

SUMMARY:
BCG has marked immune stimulatory effects in both animal and human studies and observational studies suggest that BCG is associated with a non-specific reduction in mortality in areas with high infant and child mortality. The specific objective of the study is to examine the effect of revaccination for purified protein derivative of tuberculin (PPD) reaction, scar size, morbidity and mortality in a randomised prospective study of revaccination versus no revaccination among children 19 months of age in Guinea-Bissau. The hypothesis is that revaccination with BCG reduces childhood mortality after 19 months of age by 30%.

DETAILED DESCRIPTION:
Examine in a randomised trial whether revaccination with BCG reduces childhood mortality after 19 months of age by 30%.

Criteria for verification: 3,000 children aged 1½ year enrolled and followed for an average of 3 years; information on potential adverse events among children with a positive PPD reaction; assessment of parasitaemia after revaccination; assessment of the tuberculin response and scar-formation after revaccination; and assessment of all-cause mortality during the period of follow-up.

Following consent to participate, children will be assessed for BCG scar and tuberculin reaction at 18-19 months of age. Subsequently, the children will be invited to a clinical examination at one of the health centres. The study will be explained again to the mother, and if she accepts to participate, she will draw a randomisation number deciding whether the child will be revaccinated or not. The BCG vaccine given will be the standard dose of 0.1 ml as recommended by WHO in this age group. In the beginning of the study, a group of 800 revaccinated and not revaccinated children will be followed weekly for two months to monitor morbidity and possible adverse effects of the vaccination. It is not expected that Koch like reactions will be common in this age group. However, should there be too many adverse reactions among children with a positive tuberculin test, only tuberculin negative children will be included in the continuation of the trial.

Two months after inclusion, the children will have another tuberculin test to examine changes in tuberculin reaction. At the same time, scar-size will be measured. In the initial phase of the project, a finger-prick blood sample will be collected from 1000 children to examine whether BCG boosting/no boosting have had an effect on the prevalence of malaria parasitaemia and the level of measles antibodies. Children with malaria will be treated and children with non-protective levels of measles antibodies will be offered revaccination with measles vaccine. In a group of children, samples will be collected both before and after BCG revaccination/no revaccination to measure changes in cytokine profile. Children with a large PPD reaction (> 15mm) will be followed in a similar way as the other children as this may reflect immune stimulation from exposure to natural TB. The studies of morbidity and immunological changes will be done both in the dry and the rainy seasons. The children will be followed for hospitalisations and mortality to 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* No overt illness

Exclusion Criteria:

* PPD reaction >15mm

Ages: 19 Months to 24 Months | Sex: All
Age Groups: Child
Enrollment: 2871 (Actual)
Dates: Start 2002-07; Primary Completion 2006-05 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Mortality till 5 years of age
Hospitalisations till 5 years of age
Adverse effects within 12 months after intervention

SECONDARY OUTCOMES:
Tuberculin reaction 2 months after intervention
Scar reaction 2 months after intervention
Malaria morbidity/parasitaemia within 12 months after intervention
Assessment of antibody and cellular immune responses 18 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Apartado 861, Bissau, Guinea-Bissau